CLINICAL TRIAL: NCT07077551
Title: NALIRIFOX as Second-Line Chemotherapy in Extrapulmonary High-grade Neuroendocrine Neoplasms: a Prospective, Single-center, Single-arm Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0428
Record Dates: First submitted 2025-06-27; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-04

CONDITIONS: NENS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NALIRIFOX (Experimental): NALIRIFOX
  Interventions: Drug: NALIRIFOX

INTERVENTIONS:
Drug: NALIRIFOX — A cycle will be repeated every 14 days. G-CSF prophylaxis will be allowed after each cycle. Patients will undergo re-staging studies every 8 weeks. Patients will receive up to 12 cycles during the study. Additional cycles will be determined per investigators' discretion.

SUMMARY:
High-grade neuroendocrine neoplasms (NENs) comprise both well-differentiated grade 3 neuroendocrine tumors (G3 NETs) and poorly differentiated neuroendocrine carcinomas (NECs). Mixed neuroendocrine-non-neuroendocrine neoplasms (MiNENs) nearly always include poorly differentiated NEC as the neuroendocrine component. Liposomal irinotecan hydrochloride and NALIRIFOX (liposomal irinotecan hydrochloride with fluorouracil and oxaliplatin) obtained a significant breakthrough in pancreatic cancer treatment. While the efficacy and safety of NALIRIFOX has never been investigated in patients with extrapulmonary high-grade NENs.

Investigators conducted a two-stage, prospective, single-center, single-arm trial which enrolled patients with extrapulmonary advanced high-grade NENs who failure of first-line treatment. The primary endpoint is 6-moth disease-free survival. The second endpoint is disease control rate. Investigators will enroll 12 patients in first stage. If more than 6 patients reach 6-moth disease-free survival, the research enters the next stage.

Investigators will enroll 28 patients in total, and if more than 19 patients reach the primary endpoint, investigators will further design the phase III clinical trail.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written Informed Consent Form to voluntarily enroll in this study.
2. Men or women aged 18-75.
3. Histologically or cytologically confirmed metastatic neuroendocrine carcinoma, neuroendocrine tumour G3 or mixed neuroendocrine-non-neuroendocrine tumour (neuroendocrine component >30%)
4. Patients who have failed one previous systemic treatment.
5. ECOG PS score of 0 or 1.
6. Life expectancy is at least 3 months.
7. The investigator assessed the presence of measurable lesions at baseline by imaging (according to RECIST 1.1), and measurable lesions should not have received local treatment such as radiotherapy (lesions located within the area of previous radiotherapy may also be selected as target lesions if progression is confirmed to have occurred).
8. Function of vital organs in accordance with the following requirements (no blood components, cell growth factor corrective therapy with any medication is permitted within 14 days prior to the first use of the study drug); ① Absolute neutrophil count (ANC) ≥1.5×109/L

   ② Platelets ≥ 100 x 109/L;

   ③ Haemoglobin ≥ 8g/dL;

   ④ Total bilirubin ≤ 1.5 × ULN; ALT, AST ≤ 2.5 × ULN, and if liver metastases are present, ALT, AST ≤ 5 × ULN;

   ⑤ Serum creatinine ≤ 1.5 × ULN or creatinine clearance > 60 mL/min (Cockcroft-Gault);
9. Female subjects of childbearing potential are required to have a negative serum pregnancy test within 72 hours prior to initiation of trial drug administration and to use effective contraception (e.g., IUD, birth control pills, or condoms) during the trial period and for at least 3 months after the last dose; male subjects whose partner is a female of childbearing potential are required to use effective contraception during the trial period and for at least 3 months after the last dose. For male subjects whose partners are women of childbearing potential

Exclusion Criteria:

1. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects who have been previously treated for brain metastases may participate in treatment provided they have stable brain metastases and have not been treated for brain metastases with steroids for at least 28 days prior to study entry. This exception does not include carcinomatous meningitis, as patients with carcinomatous meningitis are excluded regardless of clinical stability;
2. Major surgery, open biopsy or severe trauma 28 days prior to first dose;
3. Prior history of allergy to fluorouracil or irinotecan;
4. Have high blood pressure that is not well controlled by antihypertensive medication (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg)
5. Subjects with uncontrolled cardiovascular clinical conditions or disease, including but not limited to: e.g., (1) NYHA class II or higher heart failure (2) unstable angina (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmia not controlled without or with clinical intervention
6. Have experienced clinically significant bleeding symptoms or have a definite tendency to bleed within 3 months prior to the first dose, e.g. peptic haemorrhage, haemorrhagic gastric ulcer or have vasculitis;
7. Arterial/venous thrombotic events such as cerebrovascular accidents (including temporary ischaemic attack, cerebral haemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism occurring within 6 months prior to the first dose of the drug, with superficial vein thrombosis being eligible for enrolment as determined by the investigator; and
8. There is another malignancy that is progressing or requires active treatment, with the exception of non-melanoma skin cancers and cervical cancer in situ for which potential treatment has already been undertaken;
9. Women who are pregnant or breastfeeding;
10. In the judgement of the investigator, the subject has other factors that may cause him/her to be forced to terminate the study midway, such as other serious illnesses (including psychiatric illnesses) that require comorbid treatment, severely abnormal laboratory test values, family or social factors that may affect the subject's safety or the collection of experimental data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
6-month Progression-Free Survival | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Objective Response Rate | 1 year
Disease Control Rate | 1 year
Overall Survival | 1 year
Quality of Life (QoL) assessment | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No